CLINICAL TRIAL: NCT00688103
Title: Efficacy and Safety of Etanercept in Active Rheumatoid Arthritis Despite Methotrexate Therapy in Japan
Brief Title: Efficacy and Safety of Etanercept in Active RA Despite Methotrexate Therapy in Japan
Acronym: JESMR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Japan Biological Agent Study Integrated Consortium (Network)
Responsible Party: Principal Investigator, Hideto Kameda, Professor, Toho University, Japan Biological Agent Study Integrated Consortium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Etanercept-01
Record Dates: First submitted 2008-05-25; First posted 2008-06-02 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ETN Alone (Active Comparator): etanercept (25mg, twice/week, s.c.)
  Interventions: Drug: ETN Alone
- ETN+MTX (Active Comparator): etanercept (25mg, twice/week, s.c.) combined with methotrexate (6-8mg/week)
  Interventions: Drug: ETN+MTX

INTERVENTIONS:
Drug: ETN Alone — etanercept (25 mg, twice/week, s.c.)
  Other Names: etanercept
  Arms: ETN Alone
Drug: ETN+MTX — etanercept (25 mg, twice/week, s.c.) combined with methotrexate (6-8 mg/week)
  Other Names: etanercept and methotrexate
  Arms: ETN+MTX

SUMMARY:
Multi-center, parallel-group, randomized, open control study. All patients will be selected to two treatment groups.

1. Etanercept alone treatment group (25mg, twice/week, s.c.)
2. Etanercept combined with MTX group (25mg, twice/week, s.c.+MTX 6-8mg/week)

ELIGIBILITY:
Inclusion Criteria:

* Patients had to be at least 18 years of age
* fulfilled the 1987 revised classification criteria for RA by in American College of Rheumatology (ACR)
* met the guidelines for the proper use of ETN in Japan (having at least 6 tender joints and 6 swollen joints
* either serum C-reactive protein more than 2 mg/dl or ESR no less than 28 mm at 1 hour, with adequate safety profiles)
* be ACR functional class I-III
* have been receiving MTX 6 mg/week for a minimum of 3 months at a stable dose for at least 4 weeks at the time of study enrollment

Exclusion Criteria:

* Patients who required concurrent use of prednisone (PSL) >10 mg/day, or its equivalent, were excluded from study entry
* the start of dose increment of PSL equivalents within 3 months of the study enrollment
* experience of antirheumatic therapy except for MTX and PSL equivalents
* previous treatment with ETN or any other biological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2005-06; Primary Completion 2008-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, MD, PhD, Study Chair — JBASIC
Locations (1):
- Keio University, Tokyo, Tokyo, Japan

REFERENCES:
- [Result] Kameda H, Ueki Y, Saito K, Nagaoka S, Hidaka T, Atsumi T, Tsukano M, Kasama T, Shiozawa S, Tanaka Y, Takeuchi T; Japan Biological Agent Study Integrated Consortium. Etanercept (ETN) with methotrexate (MTX) is better than ETN monotherapy in patients with active rheumatoid arthritis despite MTX therapy: a randomized trial. Mod Rheumatol. 2010 Dec;20(6):531-8. doi: 10.1007/s10165-010-0324-4. Epub 2010 Jun 24. PMID 20574649
- [Result] Kameda H, Kanbe K, Sato E, Ueki Y, Saito K, Nagaoka S, Hidaka T, Atsumi T, Tsukano M, Kasama T, Shiozawa S, Tanaka Y, Yamanaka H, Takeuchi T. Continuation of methotrexate resulted in better clinical and radiographic outcomes than discontinuation upon starting etanercept in patients with rheumatoid arthritis: 52-week results from the JESMR study. J Rheumatol. 2011 Aug;38(8):1585-92. doi: 10.3899/jrheum.110014. Epub 2011 May 15. PMID 21572151
- [Result] Kameda H, Kanbe K, Sato E, Ueki Y, Saito K, Nagaoka S, Hidaka T, Atsumi T, Tsukano M, Kasama T, Shiozawa S, Tanaka Y, Yamanaka H, Takeuchi T; Japan Biological Agent Integrated Consortium (JBASIC). A merged presentation of clinical and radiographic data using probability plots in a clinical trial, the JESMR study. Ann Rheum Dis. 2013 Feb;72(2):310-2. doi: 10.1136/annrheumdis-2012-201804. Epub 2012 Sep 12. No abstract available. PMID 22975754

RESULTS

PARTICIPANT FLOW:
Groups:
- ETN Alone: Etanercept alone treatment group (25mg, twice/week, s.c.)
- ETN+MTX: Etanercept combined with MTX group (25mg, twice/week, s.c.+MTX 6-8mg/week)
Period: Overall Study
Arm/Group | ETN Alone | ETN+MTX
Started | 74 | 77
Actually Treated | 71 | 76
Completed | 44 | 64
Not Completed | 30 | 13
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 11 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — complex reasons | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETN Alone | ETN+MTX | Total
Number analyzed (Participants) | 74 | 77 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 58 | 112
  >=65 years | 20 | 19 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.6) | 56.6 (11.1) | 57.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 62 | 127
  Male | 9 | 15 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 74 | 77 | 151

OUTCOME MEASURES:

1. Primary Outcome: EULAR Good Response
Description: EULAR good response was defined as reaching, at least, low decease activity by the disease activity score of 28 joints (DAS28) and its improvement by > 1.2. DAS28 is a quantitative composite measure of disease activity for rheumatoid arthritis, and DAS28 < 3.2 is regarded as low disease activity.
Time Frame: at 24 weeks
Measure: Number; unit: percentage of responders
Arm/Group | ETN Alone | ETN+MTX
Number analyzed (Participants) | 69 | 73
percentage of responders | 33.3 | 52.1

2. Primary Outcome: ACR50 Response Rate
Description: ACR (American College of Rheumatology) 50 response is defined by the following definition of improvement: at least 50% improvement in tender and swollen joint counts and at least 50% improvement in 3 of the 5 remaining ACR-core set measures; patient and physician global assessments, pain, disability, and an acute phase reactant (erythrocyte sedimentation rate or C-reactive protein).
Time Frame: at 24 weeks
Measure: Number; unit: percentage of responders
Arm/Group | ETN Alone | ETN+MTX
Number analyzed (Participants) | 69 | 73
percentage of responders | 47.8 | 64.4

3. Primary Outcome: Radiographic Progression Defined by Change in Van Der Heijde-modified Total Sharp Score
Description: The van der Heijde-modifiedtotal Sharp score is the sum of scores for erosions and joint space narrowing. The minimum and maximum total scores are 0 and 448, respectively. The maximum number of erosions is 160 in the hands and 120 in the feet; and the maximum scores for joint space narrowing are 120 and 48, respectively.
  Erosions are scored 1 for a discrete interruption of the cortical surface, and scored 2-5 for a larger defect according to the surface area of the joint involved. Notably, the maximum erosion score in each joint in hands is 5, while it is 10 in the feet.
  For joint space narrowing, 0=normal; 1=focal or doubtful; 2=general, <50% of the original joint space; 3=general, >50% of the original joint space or subluxation; 4=ankylosis.
Time Frame: at 52 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ETN Alone | ETN+MTX
Number analyzed (Participants) | 53 | 68
units on a scale | 3.6 (10.4) | 0.8 (6.4)

ADVERSE EVENTS:
Arm/Group | ETN Alone | ETN+MTX
Serious Adverse Events (participants affected / at risk) | 2/71 | 9/76
Other Adverse Events (participants affected / at risk) | 34/71 | 39/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETN Alone (N=71) | ETN+MTX (N=76)
bone fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2)
congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1)
brain hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
mammary carcinoma (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETN Alone (N=71) | ETN+MTX (N=76)
upper airway viral infection (Infections and infestations) | 29 (55) | 33 (55)
gastroentelitis (Gastrointestinal disorders) | 7 (7) | 8 (8)
injection site reaction (General disorders) | 16 (16) | 9 (9)
rash (Skin and subcutaneous tissue disorders) | 19 (19) | 8 (8)
mild injury (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
headache (Nervous system disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No